CLINICAL TRIAL: NCT05167578
Title: Identifying Reasons for Non-adherence in Patients With Multi-morbidity: A Protocol for Prospective Observational Study in Primary Care
Brief Title: Identifying Reasons for Non-adherence in Patients With Multi-morbidity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Kirsi Kvarnström, Senior pharmacist in charge, Helsinki University Central Hospital
Other Study IDs: HUS/1037/2020; VD/4977/13.00.00/2020 (Other: The Institutional Review Board Vantaa)
Record Dates: First submitted 2021-11-19; First posted 2021-12-22 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Medication Adherence; Medication Nonadherence; Chronic Disease
Keywords: medication adherence; nonadherence; self-management; chronic disease; multimorbidity; primary care; medication reconciliation; pharmacist; public health
MeSH Terms: conditions — Medication Adherence; Chronic Disease | interventions — Medication Reconciliation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with multimorbidity: Patients with multimorbidity who visit the public health centres in Vantaa, Southern Finland
  Interventions: Behavioral: Medication reconciliation

INTERVENTIONS:
Behavioral: Medication reconciliation — A pharmacist will go through all medicines physicians have prescribed, over-the-counter medicines (OTC) and food supplements one by one to assess the actual medicine used by the patient. If a pharmacist identifies medication discrepancies between physician's prescriptions and patient's self-reported use of medicine during the medication reconciliation, she/he will find out the patients' reasons for adjusting the medication.

SUMMARY:
The study will be carried out during pharmacist-conducted medication reconciliation. The pharmacist will ask how the patient has been taking the prescribed medicines and whether any over-the-counter medicines and food supplements have been used for self-medication. The data will be analyzed for descriptive statistics to identify 1) the number of discrepancies between the physician's prescription orders and the patient's self-reported use of the medicines, 2) what kind of discrepancies there are, and 3) which of them negatively influence patients' medicine taking.

DETAILED DESCRIPTION:
This study aims to identify patient-reported reasons for medication non-adherence during pharmacist-led medication reconciliation in primary care. The investigators will examine medication discrepancies between physicians' prescription orders and patients' self-reported medication use, which medicines patients most often use against physician's order, and the reasons for the variant use of medicines. Additionally, the investigators will study the correlation between medication discrepancies and the number of medicines the patient uses. The investigators also aim to investigate which medicines can be classified as high-risk medicines for non-adherence.

The research method will contain a pharmacist-conducted medication reconciliation including a patient interview in a 30-minute appointment. Physicians, nurses, and pharmacists identify patients who are eligible for this study. The study will include 250 patients who visit the public health centres in Vantaa, Southern Finland.

Medication reconciliation will take place at the admission to the health centre, usually before physicians' appointments. A pharmacist will go through all medicines physicians have prescribed, over-the-counter medicines (OTC) and food supplements one by one to assess the actual medicine used by the patient. If a pharmacist identifies medication discrepancies between physician's prescriptions and patient's self-reported use of medicine during the medication reconciliation, she/he will find out the patients' reasons for adjusting the medication. Based on this process pharmacist formulates the updated medication list, including clinically appropriate over-the-counter medicines (OTC medicines) in the patient record system Apotti, where the physician will once more make sure that everything is in order. The pharmacist will advise the patient to clarify the possible misunderstandings or concerns toward medications and motivate the patient to use the medication as prescribed. The outcome of the discussion is documented.

The data will be analyzed by descriptive statistical analysis. The patients' reported reasons for medication discrepancies will be analyzed quantitatively, and central themes and subthemes will be classified. The risk ratio will be identified, i.e., the relative risk among the number of medicines and medication discrepancies. The investigators will compare the total number of patients' medicine, including non-prescription medicine, to medicine the patient is using differently as prescribed and calculate the possible comparative risk adjusting the medicine with the number of prescribed medicines. The investigators will also identify the high-risk medications for non-adherence. The investigators will analyze patients' need for information on medicines as the patient receives guidance and encouragement when the pharmacist identifies discrepancies. The data will be analyzed using IBM SPSS Statistics 26 software.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multimorbidity
* Patients with ≥5 prescription medicines
* Finnish speaking
* Living at home and managing daily life independently
* Willingness to take part and sign the informed consent

Exclusion Criteria:

* Patients not understand Finnish
* Diagnosed Alzheimer or another memory disorder
* Need help to manage daily life
* End of life care

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic conditions and multiple medication who visit the public health centres in Vantaa, Southern Finland
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Medication discrepancy | Through study completion, an average of 3 months
  Comparison of actual use of medicines versus prescribed medicines

SECONDARY OUTCOMES:
The groups of medicines | Through study completion, an average of 3 months
  The medicines that are used differently as prescribes are classified in anatomical therapeutic chemical groups
The reason for non-adherence | Through study completion, an average of 3 months
  Patient reported reasons for not taking medicines as prescribed
The effectiveness of medication information | Through study completion, an average of 3 months
  Will the patient consider taking the medication as prescribed after the discussion with the pharmacist

CONTACTS AND LOCATIONS:
Overall Officials: Marja Airaksinen, PhD Pharm, Study Director
Locations (1):
- Vantaa healthcare and social services, Vantaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided
All data relevant to the study will be included in the article or uploaded as supplementary information. The data does not include patient identifiable data.

REFERENCES:
- [Derived] Kvarnstrom K, Westerholm A, Airaksinen MS, Liira H. Why medicines are used differently from prescribed: a protocol for a prospective patient-oriented observational case study to investigate reasons for non-adherence in primary care. BMJ Open. 2022 Dec 22;12(12):e065363. doi: 10.1136/bmjopen-2022-065363. PMID 36549723